CLINICAL TRIAL: NCT00464386
Title: Continuous Glucose Monitors (CGM) Versus Point-of-Care (POC) Glucometers in the Intensive Care Unit (ICU)
Brief Title: Continuous Glucose Monitoring (POC) in the ICU
Acronym: POC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study device required infeasible modifications. No patients received device.
Sponsor: United States Army Institute of Surgical Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-06-011
Record Dates: First submitted 2007-04-20; First posted 2007-04-23 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2015-02

CONDITIONS: Burns; Trauma
Keywords: Severe burns; Severe Trauma; Closed loop insulin; continuous glucose monitoring
MeSH Terms: conditions — Burns; Wounds and Injuries | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- POC Glucose Testing (No Intervention): Hourly blood glucose monitoring with point of care glucometer (i.e., current standard of care).
- Continuous Glucose Monitoring (Experimental): Continuous arterial glucose monitoring with Guardian sensor + hourly blood glucose monitoring with point of care glucometer (i.e., current standard of care).
  Interventions: Device: Continuous Glucose Monitoring

INTERVENTIONS:
Device: Continuous Glucose Monitoring — measure glucose levels on burn patients
  Other Names: Guardian continuous glucose monitor
  Arms: Continuous Glucose Monitoring

SUMMARY:
The purpose of this study is to prospectively evaluate whether the addition of continuous glucose monitoring to point-of-care (POC) glucometer monitoring improves glucose control.

DETAILED DESCRIPTION:
Severe burns and traumatic injury can be associated with protracted illness and prolonged ICU course. The beneficial effects of strict serum glucose control in critically ill surgical patients have been demonstrated. Continuous glucose monitors may improve glucose control by providing close to real-time glucose measurements, giving the critical care team the ability to react to trends before hypo- or hyperglycemia is reached. These improvements may decrease the morbidity and mortality associated with severe thermal injury, thereby minimizing hospital stay and recovery. Burned and injured soldiers, airmen, sailors, and marines may return to duty in a more expeditious fashion, or at minimum, enjoy a better quality of life after discharge from the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* remain 1 week in an ICU
* 18-72 years old
* severe trauma or thermal injury greater than 20% TBSA burn

Exclusion Criteria:

* cerebral arterial injury
* myocardial infarction
* pre-existing renal failure or liver failure
* history of hypoglycemia
* history or high risk of seizures
* pregnancy

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-09; Primary Completion 2009-02 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To prospectively evaluate the reliability of continuous glucose monitors and the advisability of their use in patients with severe trauma and or thermal injury. | 90 days

SECONDARY OUTCOMES:
To investigate whether the use of continuous glucose monitoring systems in the ICU results in better glucose control. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Heather Pidcoke, MD, Principal Investigator — US Army Institute of Surgical Research
Locations (1):
- US Army Institute of Surgical Research, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kerr D. Continuous blood glucose monitoring: detection and prevention of hypoglycaemia. Int J Clin Pract Suppl. 2001 Sep;(123):43-6. PMID 11594298